CLINICAL TRIAL: NCT03633747
Title: Efficacy Evaluation of Propranolol Treatment of Hepatic Hemangioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Limited efficacy
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU-Y2018-059
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2018-08

CONDITIONS: Hemangioma Liver
Keywords: hepatic hemangioma; propranolol
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- propranolol (Experimental): Propranolol hydrochloride tablets were taken orally three times a day at an initial dose of 30 mg/day, doubled one week later until the daily dose was 1.5 mg/kg. If the dose was unable to increase due to side effects, the maximum dose tolerable was maintained for 6 months.
  Interventions: Drug: Propranolol Hydrochloride

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Oral propranolol hydrochloride tablets are administration for 6 months at dose of 1.5 mg/kg or the maximum dose tolerable.

SUMMARY:
Hepatic hemangioma is one of the most common benign tumor of the liver. Although the overall prognosis is good, active interventions are still needed in high-risk patients. Without specific drugs, the main treatment methods include surgical treatments, interventional therapies and radiotherapies. Effective medical treatments are needed urgently. Propranolol has achieved good results in infantile Facial/hepatic hemangioma, and shows some effectiveness in adult hemangioma. Here, investigators intend to evaluate the therapeutic effect of propranolol in adult hepatic hemangioma.

DETAILED DESCRIPTION:
In view of the lack of medical treatment for hepatic hemangioma, investigators chose hemangioma patients with a diameter of 5-10 cm and no significant risk of rupture, or those with surgical indications but rejected of surgical, interventional/radiological interventions. After confirmation of no high risk for drugs, oral propranolol was given. The tumor size, objective remission rate, disease control rate, drugs related side effects and other endpoints events were recorded and analyzed, to assess the propranolol could or couldn't effectively control the progress of hepatic hemangioma.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age.
* Hemangioma with a diameter of 5-10 cm, no clinical symptoms, no obvious risk of hemangioma rupture and bleeding, no obvious symptoms of tumor compression, and excluding malignant diseases; or hemangioma without surgical indications but have a strong willingness to treat; compliance with treatment indications, but refuse surgical, interventional or radiotherapy radiative interventions.
* No other beta receptor modulators (activation or blockade of beta receptor signaling) were given during the previous six months.
* Eastern Cooperative Oncology Group score 0-2 points.

Exclusion Criteria:

* Liver lesions with other malignant tumors or hepatic hemangiomas are not clearly diagnosed or have other undefined features.
* Hepatic hemangioma requires surgical or radiological intervention within a limited period of time, otherwise there may be a greater risk.
* Beta receptor modulator therapy is required for cardiovascular and other diseases within six months.
* Previous cardiovascular or cerebrovascular events or with high risk of cardiovascular and cerebrovascular events.
* Suffering from severe liver diseases such as severe cirrhosis, hepatic adenoma, liver dysfunction and so on.
* Post liver transplantation.
* Heart rate < 60 beats/min, blood pressure < 100/60 mmHg, orthostatic hypotension, cardiac insufficiency or severe cardiovascular disease (moderate to severe hypertension, coronary atherosclerotic heart disease, severe or acute heart failure, II-III atrioventricular block, ventricular tachycardia, cardiogenic shock, Raynaud syndrome or other peripheral vascular diseases).
* Severe pulmonary diseases (such as bronchial asthma, emphysema), severe hematological diseases (such as agranulocytosis, thrombocytopenia), severe mental disorders (such as depression), severe thyroid diseases (hypothyroidism, hormone replacement therapy after thyroidectomy), diabetes mellitus need to be controlled by drugs. Severe kidney disease (such as nephrotic syndrome, glomerulonephritis, renal insufficiency).
* Others: history of drug allergy, pregnancy or breast-feeding, other malignant tumors in the past five years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Tumor size | 6 months after treatment
  Evaluating maximum diameter obtained by contrast-enhanced CT scanning

SECONDARY OUTCOMES:
Objective response rate | 6 months after treatment
  Percentage of patients whose cancer shrinks or disappears after treatment

OTHER OUTCOMES:
Disease control rate | 6 months after treatment
  Percentage of patients whose cancer doesn't progress after treatment
Vascular endothelial growth factor | 6 months after treatment
  Level of serum Vascular endothelial growth factor
Common Toxicity Criteria for Adverse Effects | 6 months after treatment
  According to Common Toxicity Criteria for Adverse Effects version 4

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided